CLINICAL TRIAL: NCT06523621
Title: Nivolumab As An Adjunctive Therapy In Relapsed Refractory Multiple Myeloma Patients With Sub-Optimal Response To Idecabtagene Vicleucel
Brief Title: Nivolumab in Multiple Myeloma Patients After Idecabtagene Vicleucel
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB0011836; LCI-PCD-RRMM-NIVO-001 (Other: AHWFBCCC); Pro00081644 (Other: Advarra IRB)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Plasma Cell Disease; CAR-T
MeSH Terms: conditions — Multiple Myeloma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Nivolumab
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — 2 cycles of nivolumab at a dose of 480 mg given over approximately 30-minutes intravenously on Day 1 of each treatment cycle
  Other Names: Opdivo

SUMMARY:
This study is designed to evaluate if treatment with adjuvant nivolumab improves depth of response in patients with relapsed refractory multiple myeloma (RRMM) who achieve a less-than-ideal response to idecaptagene vicleucel.

DETAILED DESCRIPTION:
This is a single arm, two-stage, Phase II of adjuvant nivolumab in patients with RRMM treated with at least 2 prior lines of therapy and are refractory to or intolerant of at least one proteasome inhibitor (PI), one immunomodulatory agent (IMiD), and one anti-CD38 antibody who achieved a sub-optimal response (defined as a VGPR, PR, MR, or SD by IMWG 2016 criteria) to treatment with idecabtagene vicleucel.

This study will determine best overall response after 2 cycles of adjuvant nivolumab given every 4 weeks in patient who achieve a sub-optimal response to ide-celon restaging studies ~30 days after infusion. The Investigators will also evaluate for changes in CAR-T cell expansion, persistence of CAR-T cells, and additional toxicity compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information signed by the participant or his/her legally authorized representative
2. Age ≥ 18 years at the time of consent
3. ECOG Performance Status (PS) of ≤ 1 at the time of enrollment. PS must be evaluated within 14 days prior to enrollment.
4. Measurable disease according to IMWG 2016 criteria present within 28 days prior to ide-cel infusion. Note that patients will NOT be required to have measurable disease at time of enrollment. Measurable disease is defined as:

   1. Serum M-protein ≥1 g/dL (> 0.5 g/dL for IgA or IgM) OR
   2. Urine M-protein ≥200 mg/24 h OR
   3. Involved free light chain (FLC) level ≥10 mg/dL provided serum FLC ratio is abnormal
5. Previous treatment with idecabtagene vicleucel according to the FDA approved US prescribing information with a response of CR/sCR, VGPR or PR by IMWG 2016 criteria evaluated no sooner than 3 weeks after idecabtagene vicleucel infusion when compared to baseline disease evaluations collected no earlier than 28 days prior to ide-cel infusion. Note: The 28-day window applies to all assessments, even if assessments were performed on different days.

   Note: Participants who received non-conforming idecabtagene vicleucel who were originally prescribed idecabtagene vicleucel according to the FDA approved label may be considered for inclusion per the investigator's discretion.
6. Participants must be enrolled no sooner than 3 weeks and no later than 6 weeks from the date of the idecabtagene vicleucel infusion.
7. Recovered from all non-hematologic reversible acute toxic effects of prior therapy (other than alopecia) to ≤ grade 1 or baseline. Participants with grade ≤ 2 treatment induced peripheral neuropathy are eligible. Participants with hematologic reversible acute toxic effects are allowed to participate if laboratory values meet eligibility parameters.
8. Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 28 days prior to enrollment. The most recent labs prior to enrollment will be used to evaluate for eligibility if labs drawn more than once during screening.
9. Females of childbearing potential (FCBP) must have a negative serum pregnancy test within 72 hours prior to enrollment. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (at least 12 consecutive months with no menses without an alternative medical cause).

   FCBP must be willing to use a highly effective contraceptive method (i.e., achieves a failure rate of <1% per year when used consistently and correctly) from the time of informed consent until 5 months after last dose of nivolumab. Contraceptive methods with low user dependency are preferable but not required (see table, adapted from: 2020_09_HMA_CTFG_Contraception_guidance_Version_1.1_updated.pdf)
10. Ability of the participant to understand and comply with study procedures for the entire length of the study, as determined by the enrolling investigator

Exclusion Criteria:

1. Diagnosis of Waldenstrom macroglobulinemia, POEMS syndrome, or amyloidosis
2. History of/or active infection listed below:

   1. Active infection requiring systemic therapy (NOTE: at discretion of investigator, participants receiving treatment for an uncomplicated urinary tract infection or localized cellulitis may be eligible.)
   2. Uncontrolled Human Immunodeficiency Virus (HIV) or hepatitis B infection. Well controlled HIV infection (as defined by an undetectable viral load) and chronic hepatitis B infection on appropriate prophylaxis can be considered per enrolling investigator discretion
   3. Active hepatitis C infection. Participants with previously treated hepatitis C infection with documented eradication of their infection will be allowed to enroll.
   4. Known history of active TB (Bacillus Tuberculosis)
3. Pregnant or breastfeeding (Note: breast milk cannot be stored for future use while the mother is being treated on study.)
4. Current evidence of active cytokine release syndrome or neurotoxicity (any grade)
5. Participants previously diagnosed with an additional malignancy must be disease-free for at least 2 years prior to enrollment. Exceptions include basal cell or squamous cell skin cancer and in situ cervical or bladder cancer.
6. Treatment with any anti-myeloma therapy or investigational drug within 30 days prior to cycle 1 day 1 of nivolumab other than ide-cel with the exception of lymphodepleting chemotherapy or steroids for ide-cel therapy. Investigational includes drugs approved for human use but not approved for the indication.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator
8. History of transplant:

   1. Autologous stem cell transplant within 12 weeks of C1D1
   2. Allogeneic stem cell transplant
   3. Solid organ transplant
9. Active known or suspected autoimmune disease. Participants with Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
10. Known history of interstitial lung disease or known history of non-infectious pneumonitis
11. Inability to take Pneumocystis jirovecii (PJP) prophylaxis (either trimethoprim-sulfamethoxazole, dapsone, or pentamidine)
12. A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of C1D1 (Note: Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease)
13. Prisoners or participants who are involuntarily incarcerated
14. Known history of myocarditis, regardless of etiology
15. Known history of allergy or hypersensitivity to study drug components
16. History of serious side effects to nivolumab or ipilimumab, as defined by the enrolling investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Depth of Response | From enrollment to best response; approximately 5 months after initiating nivolumab
  Depth of response will be determined for each participant post ide-cel with adjuvant nivolumab indicating if their best overall response is a Complete Response (CR) or stringent Complete Response (sCR). The post-ide-cel disease response assessments will be calculated relative to the participant's pre-ide-cel disease assessment parameters. Responses will be determined per IMWG 2016 response criteria.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of ide-cel administration to date of progression or death, or censored as described; assessed for approximately 4 years
  PFS is defined as the duration of time from ide-cel administration to first occurrence of either progressive disease (PD) or death (from any cause). PD will be objectively determined per IMWG 2016 criteria, where progression date is date of first assessment that identified confirmed PD. If subject died without documented PD, progression date will be death date. For surviving subjects who do not have PD, PFS will be censored at the date of last disease assessment. For subjects who received subsequent anti-cancer therapy prior to documented PD, PFS will be censored at the date of last disease assessment prior to commencement of subsequent therapy. Subjects who have an initial PFS event immediately following 2 or more consecutive missed assessments will be censored at date of last assessment prior to missed assessments.
Best Overall Response | From enrollment to best response; approximately 5 months after initiating nivolumab
  Best overall response will be determined for each participant as a categorical variable indicating the participant's best overall response achieved after treatment with nivolumab, according to IMWG 2016 response criteria. The levels for best overall response will include PD, SD, MR PR, VGPR, CR, sCR.
Duration of Response (DoR) | From date of best response to date of progression or death, or censored as described; assessed for approximately 4 years
  Duration of best response will be calculated for each participant. The duration of best response interval will begin at the first disease assessment date indicating the participant's best response. The timing for progression, death, or censoring will be determined as previously described for PFS.
Minimal Residual Disease (MRD) Negativity Rate | approximately 2 months and 5 months after enrollment
  MRD response will be determined for each participant as a binary variable indicating if the participant achieved a MRD negative status after treatment with nivolumab. MRD negative status will be separately determined at 10-5 and 10-6 sensitivity.
Overall Survival | From date of ide-cel administration to date of death, or censored as described; assessed for approximately 4 years
  OS is defined as the duration of time from ide-cel administration to the date of death from any cause. Participants who are alive or lost to follow-up at the time of the analysis will be censored at the last known date they were alive.

OTHER OUTCOMES:
Number of participants with a grade 3 or higher cytokine release syndrome event | From enrollment to 100 days after the last dose of nivolumab
  A binary variable will be determined for each participant indicating whether or not the participant experienced Grade 3 or higher treatment-emergent (regardless of causality) cytokine release syndrome (CRS) per TCT Consensus Grading during study treatment (from first dose of nivolumab until 100 days after the last dose of nivolumab).
Number of participants with a grade 3 or higher infection | From enrollment to 100 days after the last dose of nivolumab
  A binary variable will be determined for each participant indicating whether or not the participant experienced a Grade 3 or higher treatment-emergent (regardless of causality) infection, according to the NCI Common Terminology for Adverse Events version 5.0 during study treatment (from first dose of nivolumab until 100 days after the last dose of nivolumab).
Number of participants with a grade 3 or higher neurotoxicity event | From enrollment to 100 days after the last dose of nivolumab
  A binary variable will be determined for each participant indicating whether or not the participant experienced a Grade 3 or higher treatment-emergent (regardless of causality) neurotoxicity event, according to the NCI Common Terminology for Adverse Events version 5.0 during study treatment (from first dose of nivolumab until 100 days after the last dose of nivolumab). Neurotoxicity events will be investigator determined.
Number of participants with a grade 3 or higher immune-related adverse event | From enrollment to 100 days after the last dose of nivolumab
  A binary variable will be determined for each participant indicating whether or not the participant experienced a Grade 3 or higher treatment-emergent (regardless of causality) immune-related adverse event, according to the NCI Common Terminology for Adverse Events version 5.0 during study treatment (from first dose of nivolumab until 100 days after the last dose of nivolumab). Immune-related events will be confirmed by investigator.
Number of participants with a grade 4, treatment-related non-hematologic adverse event | From enrollment to 100 days after the last dose of nivolumab
  A binary variable will be determined for each participant indicating whether or not the participant experienced a treatment-related Grade 4 non-hematologic adverse event, according to the NCI Common Terminology for Adverse Events version 5.0 during study treatment (from first dose of nivolumab until 100 days after the last dose of nivolumab).
Number of participants with an on-treatment grade 5 adverse event | From enrollment to 100 days after the last dose of nivolumab
  A binary variable will be determined for each subject indicating whether or not the subject experienced a grade 5 adverse event, regardless of causality, according to the NCI Common Terminology for Adverse Events version 5.0 during study treatment (from first dose of nivolumab until 100 days after the last dose of nivolumab).
Number of participants with at least one serious adverse event | From enrollment until 100 days after last dose of study treatment
  A binary variable will be determined for each participant indicating whether or not the subject had at least one adverse event that was categorized as serious, regardless of causality. Serious is defined per the study protocol and includes events that the investigator deems serious and results in the following outcomes: death, life-threatening situation, persistent or significant disability/incapacity, requires or prolongs hospitalization, congenital anomaly/birth defect in the offspring of a study participant, suspected transmission of any infectious agent via medial product, or based upon medical judgement, may jeopardize the subject and may require medical or surgical intervention to prevent one of the afore listed outcomes from occurring.
Number of participants with at least one treatment emergent adverse event | From enrollment until 100 days after last dose of study treatment
  A binary variable will be determined for each participant indicating whether or not the subject had at least one treatment-emergent adverse event, regardless of causality. Adverse events will be categorized per NCI Common Terminology for Adverse Events version 5.0. Treatment-emergent is defined per the study protocol and includes AEs that occur after treatment start that were not present at the time of treatment start or AEs that increase in severity after treatment start if the event was present at the time of treatment start.
Number of participants with at least one grade 3 or higher treatment emergent adverse event | From enrollment until 100 days after last dose of study treatment
  A binary variable will be determined for each participant indicating whether or not the subject had at least one grade 3 or higher treatment-emergent adverse event, regardless of causality. Adverse events will be categorized per NCI Common Terminology for Adverse Events version 5.0. Treatment-emergent is defined per the study protocol and includes AEs that occur after treatment start that were not present at the time of treatment start or AEs that increase in severity after treatment start if the event was present at the time of treatment start.
Number of participants who discontinued study treatment due to adverse events | From enrollment until 100 days after last dose of study treatment
  A binary variable will be determined for each participant indicating whether or not the subject discontinued study treatment due to adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Paul, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No